CLINICAL TRIAL: NCT00191373
Title: Phase II Study of Gemcitabine and Trastuzumab Therapy in Patients With HER2 Overexpressing Metastatic Breast Cancer
Brief Title: A Trial for HER2 Positive Breast Cancer Patients With Metastatic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6133; B9E-US-S270
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-09

CONDITIONS: Breast Neoplasms; Cancer of the Breast; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Trastuzumab

INTERVENTIONS:
Drug: Gemcitabine
Drug: Trastuzumab

SUMMARY:
This phase II trial that includes Gemcitabine 1,250mg/m2 to be administered over approximately 30 minutes on days 1 and 8, every 21 days and Trastuzumab 8 mg/kg IV to be administered over 90 minutes on day 1 of the first cycle, then 6mg/kg as a 30 minute infusion administered on subsequent cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer, with stage IV disease
* Tumors tested by IHC must be 3+ positive for HER2 overexpression. Tumors tested by FISH must be positive by the specific FISH assay for genetic amplification of HER2. Tumors that are 3+ by IHC but negative by FISH assay are ineligible
* Patients must have measurable disease
* Patients may NOT have received prior chemotherapy or prior trastuzumab therapy for metastatic breast cancer.
* Patients may have received prior chemotherapy and/or hormonal therapy for early stage breast cancer, including taxane-based chemotherapy regimens. Patients may NOT have received trastuzumab in the adjuvant setting unless disease free interval from completion of trastuzumab to time of relapse is greater than 12 months.

Exclusion Criteria:

* Patients who have had prior gemcitabine chemotherapy and adjuvant trastuzumab and had less than 12- month disease free interval
* Patients with known leptomeningeal carcinomatosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2002-03; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
- Overall response rates

SECONDARY OUTCOMES:
Time to disease progression,Time to treatment failure, Overall survival, Toxicity of the combination

CONTACTS AND LOCATIONS:
Overall Officials: CALL 1-877-CTLILLY (1-877-285-4559) OR 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hot Springs, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pine Bluff, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redding, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plantation, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Voorhees Township, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Logan, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CT-LILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ogden, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morgantown, West Virginia